CLINICAL TRIAL: NCT02415179
Title: Effect of Inhaled Mometasone/Formoterol Versus Inhaled Fluticasone/Salmeterol on Peripheral Airway Function in Asthma Patients
Brief Title: Effect of Inhaled Mometasone/Formoterol Versus Inhaled Fluticasone/Salmeterol in Asthma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZS-2015
Record Dates: First submitted 2015-01-29; First posted 2015-04-14 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Asthma
Keywords: Newly diagnosed asthma; peripheral airway function
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled Mometasone/formoterol (Experimental): Inhaled Mometasone/Formoterol (100/5 microgram) 2 puffs twice daily delivered by using metered dose inhaler for 6 weeks
  Interventions: Drug: Inhaled Mometasone/formoterol
- Inhaled Fluticasone/Salmeterol (Active Comparator): Inhaled Fluticasone/Salmeterol (125/25 microgram) 2 puffs twice daily delivered by using metered dose inhaler for 6 weeks
  Interventions: Drug: Inhaled Fluticasone/Salmeterol

INTERVENTIONS:
Drug: Inhaled Mometasone/formoterol — Inhaled Mometasone/formoterol (100/5 microgram) 2 puffs twice daily via metered dose inhaler for 6 weeks
  Arms: Inhaled Mometasone/formoterol
Drug: Inhaled Fluticasone/Salmeterol — Inhaled Fluticasone/Salmeterol (125/25 microgram) 2 puffs twice daily delivered by using metered dose inhaler for 6 weeks
  Arms: Inhaled Fluticasone/Salmeterol

SUMMARY:
The purpose of this study is to investigate the effectiveness of inhaled mometasone/formoterol versus inhaled fluticasone/salmeterol on peripheral airway function in treatment of asthma.

DETAILED DESCRIPTION:
Peripheral airway dysfunction is associated with poor asthma outcome including asthma exacerbation and more symptoms. The peripheral or small airway is anatomically defined by airways with 2 mm diameter or less. Several techniques have been used for evaluating peripheral airways such as spirometry, body plethysmography, impulse oscillometry and imaging studies. Since inhaled corticosteroid is corner stone for treatment of asthma, the addition of long acting beta agonist is indicated in severe asthma with poorly controlled disease despite of high dose inhaled corticosteroid.

The inhaled corticosteroid and long acting beta agonists are available for treating asthma. There were different results in comparison studies of different inhaled corticosteroid and long acting beta agonist. These differences are related to type of inhaled formulation, potency of inhaled corticosteroid or dose and outcome measurements. The previous short term studies shown that inhaled budesonide/formoterol is superior to inhaled fluticasone/salmeterol combination for reducing of peripheral airway resistance measured by impulse oscillometry. However, the active drug was delivered by using dry powder inhaler. There is no direct comparison between inhaled mometasone/formoterol and inhaled fluticasone/salmeterol administered using metered dose inhalers. For these reasons, we conduct the open label study comparing the effect of two inhaled corticosteroid and long acting beta agonist in newly diagnosed asthma who are eligible for being treated with such combination therapies.

Eligible patients who have clinically diagnosed asthma requiring treatment with combined inhaled corticosteroid and long acting beta agonist according to Global Initiative for Asthma (GINA) guideline. The patients will be randomized to receive either inhaled mometasone/formoterol (100/5 microgram) 2 puffs twice daily or inhaled fluticasone/salmeterol (125/25 microgram) 2 puffs twice daily administered using metered dose inhalers.

The primary outcome is peripheral airway function measured by airway resistance at 5 and 20 Hz frequency from impulse oscillometry. The secondary outcome are peak expiratory flow rate, forced expiratory flow at 1 second, forced vital capacity, forced expiratory flow at 25-75% of vital capacity (FEF25-75%) measured by spirometry, residual volume per total lung capacity ratio measured by body plethysmography ,asthma control test score and asthma control questionaire-7 version. All outcome are measured at baseline and 6-week post treatments in both arms.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed asthma according to Global Initiative for Asthma (GINA) guideline 2014 without previous treatment of inhaled corticosteroid and long acting beta agonists
2. Patients with asthma symptoms of most days or wake up due to asthma one time per week or more
3. Patients with the presence of any risk factors of asthma according to Global Initiative for Asthma (GINA) guideline 2014
4. Patients with severe uncontrolled asthma
5. Patients with previous asthma exacerbation
6. Patients give consent form

Exclusion Criteria:

1. Patients with contra-indication for performing spirometry according to American Thoracic Society (ATS) and European Respiratory Society (ERS) statement of standardization for spirometry
2. Patients refuse to participate study -

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Peripheral airway function measured by impulse oscillometry | 6 weeks
  The measuring of airway resistance at 5 and 20 Hz

SECONDARY OUTCOMES:
Peak expiratory flow rate | 6 weeks
  Peak expiratory flow rate
Forced expiratory volume at 1 second | 6 weeks
  Forced expiratory volume at 1 second
Forced vital capacity | 6 weeks
  Forced vital capacity
Forced expiratory flow rate at 25-75% of vital capacity | 6 weeks
  Forced expiratory flow rate at 25-75% of vital capacity
Asthma control test score | 6 weeks
  Asthma control test score
Asthma control questionnaire-7 version | 6 weeks
  Asthma control questionnaire-7 version

CONTACTS AND LOCATIONS:
Overall Officials: Tananchai Petnak, M.D., Principal Investigator — Pulmonary and critical care, Department of Medicine, Ramathibodi Hospital, Mahidol University; Theerasuk Kawamatawong, M.D., Principal Investigator — Pulmonary and critical care, Department of Medicine, Ramathibodi Hospital, Mahidol University; Prapaporn Pornsuriyasak, M.D., Principal Investigator — Pulmonary and critical care, Department of Medicine, Ramathibodi Hospital, Mahidol University; Viboon Boonsarngsuk, M.D., Principal Investigator — Pulmonary and critical care, Department of Medicine, Ramathibodi Hospital, Mahidol University; Naparat Amornputtisathaporn, M.D., Principal Investigator — Pulmonary and critical care, Department of Medicine, Ramathibodi Hospital, Mahidol University
Locations (1):
- Faculty of Medicine, Ramathibodi Hospital, Bangkok, Thailand

REFERENCES:
- [Background] Kraft M, Pak J, Martin RJ, Kaminsky D, Irvin CG. Distal lung dysfunction at night in nocturnal asthma. Am J Respir Crit Care Med. 2001 Jun;163(7):1551-6. doi: 10.1164/ajrccm.163.7.2008013. PMID 11401872
- [Background] Martin RJ. Therapeutic significance of distal airway inflammation in asthma. J Allergy Clin Immunol. 2002 Feb;109(2 Suppl):S447-60. doi: 10.1067/mai.2002.121409. PMID 11842317
- [Background] Usmani OS, Biddiscombe MF, Barnes PJ. Regional lung deposition and bronchodilator response as a function of beta2-agonist particle size. Am J Respir Crit Care Med. 2005 Dec 15;172(12):1497-504. doi: 10.1164/rccm.200410-1414OC. Epub 2005 Sep 28. PMID 16192448
- [Background] Meltzer EO, Kuna P, Nolte H, Nayak AS, Laforce C; P04073 Study Investigators. Mometasone furoate/formoterol reduces asthma deteriorations and improves lung function. Eur Respir J. 2012 Feb;39(2):279-89. doi: 10.1183/09031936.00020310. Epub 2011 Aug 4. PMID 21828036
- [Background] Kirsten AM, Watz H, Brindicci C, Piccinno A, Magnussen H. Effects of beclomethason/formoterol and budesonide/formoterol fixed combinations on lung function and airway inflammation in patients with mild to moderate asthma--an exploratory study. Pulm Pharmacol Ther. 2015 Apr;31:79-84. doi: 10.1016/j.pupt.2014.08.007. Epub 2014 Sep 4. PMID 25194884
- [Background] Bernstein DI, Hebert J, Cheema A, Murphy KR, Cherrez-Ojeda I, Matiz-Bueno CE, Kuo WL, Nolte H. Efficacy and onset of action of mometasone furoate/formoterol and fluticasone propionate/salmeterol combination treatment in subjects with persistent asthma. Allergy Asthma Clin Immunol. 2011 Dec 7;7(1):21. doi: 10.1186/1710-1492-7-21. PMID 22152089
- [Background] Hozawa S, Terada M, Hozawa M. Comparison of budesonide/formoterol Turbuhaler with fluticasone/salmeterol Diskus for treatment effects on small airway impairment and airway inflammation in patients with asthma. Pulm Pharmacol Ther. 2011 Oct;24(5):571-6. doi: 10.1016/j.pupt.2011.05.004. Epub 2011 May 23. PMID 21624490